CLINICAL TRIAL: NCT04656314
Title: Renal Functional Magnetic Resonance Imaging in Healthy Persons - Reproducibility and Impact of Stress
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 76158
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants aged 18 to 40: 3 identical functional MRI scans. Blood samples to quantify level of physiological stress are taken before and after each scan.
  Interventions: Diagnostic Test: Functional MRI scan
- Healthy participants aged 60 and above: 3 identical functional MRI scans. Blood samples to quantify level of physiological stress are taken before and after each scan.
  Interventions: Diagnostic Test: Functional MRI scan

INTERVENTIONS:
Diagnostic Test: Functional MRI scan — Functional MRI scan: Phase contrast, BOLD, Arterial Spin Labeling, Diffusion weighted MRI, T1 mapping, T1rho mapping

SUMMARY:
The main purpose of the study is to describe the applicability and reproducibility of functional MRI scans of the kidneys in healthy participants. Furthermore, the study examines to what extent physiological stress caused by lying in a scanner affects the renal perfusion and thus the reproducibility

DETAILED DESCRIPTION:
2 groups of 10 healthy participants each are included. 1 group aged 18 to 40 and a group of participants above 60 years of age.

The functional MRI sequences are performed consecutively in a protocol set up on a 1,5 T MRI scanner.

In totl, 3 identical scans are being performed. 2 scans on day 1 followed by another scan 1-2 weeks later. Before and after each scan, cortisol and copeptin is controlled in a blood sample to quantify the level of physiological stress.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40
* Age of 60 or above

Exclusion Criteria:

* Known kidney or cardiovascular disease
* Medicine of any kind, that must be taken on days of scanning
* MRi incompatible implants or other contraindications to MRi
* Claustrophobia
* Not being able to lie still in an hour
* Body weight above 110 kg or waist circumference above 95 cm
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
Reproducibility | Results from scans performed with an interval of 1 to 2 weeks are compared
  Reproducibility as a coefficient of variation
Physiological stress | Results from scans performed with an interval of 1 to 2 weeks are compared
  Quantified by level of cortisol and copeptin in blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: Undecided